CLINICAL TRIAL: NCT01314534
Title: French Kabuki Syndrome Network. Epidemiology, Management of Patients and Research by Array-CGH
Acronym: Kabuki
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 07-090 / P070130; IDRCB 2007-A00912-51 (Other: AFSSAPS)
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Kabuki Syndrome
Keywords: Kabuki syndrome; Genetic; CGH-array
MeSH Terms: conditions — Kabuki syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Create a census for the duration of the search for French patients with SK

* determining epidemiological and morphological parameters,
* determine the true frequency of clinical symptoms and identify new ones,
* identify complications of the disease to improve the care of patients in the hope of a better prognosis of the disease and
* performing a radiological study by Voxel based morphometry MRI type (N. BODDAERT, HOPITAL Necker-Enfants Malades, Paris)

Perform genetic research to identify the genetic bases of SK using CGH-array (Comparative Genomic Hybridization )

DETAILED DESCRIPTION:
Kabuki syndrome (KS) is a rare syndrome, sporadic dominant condition with a frequency of 1 / 35000 (between 20 and 25 new children by year in France). Five cardinal criteria have been described for this diagnosis: postnatal growth retardation, mild to moderate mental retardation, skeletal abnormalities, dermatoglyphic abnormalities and characteristic facial dysmorphism. Moreover, a large number of other symptoms are described in KS. Each year, new symptoms are reported in the international literature but without their true frequency or recommendations for the management of patients. However, these criteria are not always present in patients and there is no major or minor criteria for establishing the diagnosis. Nowadays, knowledge of this syndrome is still very fragmentary. At the date of the creation of the network, no molecular basis has been identified for the SK.

We propose to create a national network of geneticists including 18 centers labeled "developmental defects" and / or mental retardation in France gathered in Federation Development Centers labeled anomalies (the FECLAD, Head, Professor A VERLOES, Hospital Robert Debré, Paris). We will also rely on Kabuki Syndrome Association that gives us logistical support with families.

The objective of the French Kabuki syndrome network of (FKSN) is to establish a national network to:

1. create a census for the duration of the search for French patients with SK (expected number of patients = 110) for

   * determining epidemiological and morphological parameters,
   * determine the true frequency of clinical symptoms and identify new ones,
   * identify complications of the disease to improve the care of patients in the hope of a better prognosis of the disease and
   * performing a radiological study by Voxel based morphometry MRI type (N. BODDAERT, HOPITAL Necker-Enfants Malades, Paris)

   And
2. perform genetic research to identify the genetic bases of SK using CGH-array (Comparative Genomic Hybridization ).

The RFSK will be responsible for recruiting and evaluating patients with SK, the data collection and informed consent from patients for participation in the project and the establishment of rules for management of patients.

We will also perform MRI Voxel based morphometry in a small cohort of 10 patients aged 8 to 15 years to identify abnormal brain region distribution in patients with abnormal SK. The cohort of patients will be paired with SK-age compared to a historical control cohort and the cohort of patients with SK will be in uniform after the completion of IQ-type test WISC-Wechsler Intelligence Scale for Children-IV (tests performed routinely in all center for each patient).

The RFSK will also be responsible for collecting blood samples with informed consent of patients for molecular studies. These samples will be centralized in the CRB's Hospital Necker-Enfants Malades (Head: Prof. CORINNE ANTIGNAC) for the establishment of lymphoblastoid lines and bases of white blood cells.

Because of the lack of standard methodology of studies of candidate genes relevant in the rare disease, we will take genetic research, using these samples to identify the genetic basis of KS using array CGH high density (44000 clones) on an AGILENT platform (Dr. D SANLAVILLE, Lyon). This research, already used successfully in other sporadic dominant rare diseases (such as CHARGE syndrome), we may help to identify an anomaly INFRACYTOGENETIQUE to locate the gene responsible for SK.

ELIGIBILITY:
Inclusion criteria :

* diagnosis based on the decision of National Network of Geneticists
* signed informed consent by the 2 parents
* signed informed consent by the 2 parents to participate to molecular study

Exclusion criteria :

* absence of social insurance
* refusal of the patient and /or parents to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cross-sectional multicenter exploratory and observational study
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2008-09; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Determining epidemiological and morphological parameters | 2 YEARS
  * determining epidemiological and morphological parameters,
  * determine the true frequency of clinical symptoms and identify new ones,
  * identify complications of the disease to improve the care of patients in the hope of a better prognosis of the disease
  * performing a radiological study by Voxel based morphometry MRI type

SECONDARY OUTCOMES:
Perform genetic research to identify the genetic bases of SK using CGH-array | 2 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas LYONNET, PU-PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Department of Genetic, Necker Hospital, Paris, France